CLINICAL TRIAL: NCT07054437
Title: Video-based Assessment of Preschool Children's Gross Motor Development for Early Intervention Screening
Brief Title: Video-based Assessment of Preschool Children's Gross Motor Development
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: 2501160032
Record Dates: First submitted 2025-06-10; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Gross Motor Development Delay
Keywords: artificial intelligence; machine learning; neural networks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gross Motor Development Screening Tool — This intervention is an automated gross motor development screening tool specifically designed for independently walking children aged one to six years old in Taiwan. What sets it apart is its use of artificial intelligence (AI) algorithms to analyze motion data, enabling early identification of potential gross motor developmental delays.
  Unlike traditional methods that rely on manual, visual observation and subjective recording by healthcare professionals, this tool aims to significantly reduce assessment time and human resource costs. Furthermore, its automated nature makes it uniquely suited for telemedicine applications, allowing for remote screenings and overcoming geographical barriers to access early intervention services. The tool will be developed and validated against established developmental norms relevant to the Taiwanese population.

SUMMARY:
Artificial intelligence (AI) is currently one of the global focal points for industrial development, with its applications in healthcare steadily increasing, such as in disease prediction, image diagnosis, and drug development. AI assists healthcare professionals in clinical decision-making by training relevant models through algorithms, thereby enhancing medical efficiency and quality.

Currently, standardized tools are used in clinical settings to screen and assess various aspects of child development. Children's motor development levels are determined by comparing their performance against established norms. However, the current assessment methods primarily rely on on-site visual observation and recording by evaluators, which demands significant time and human resources.

This research aims to establish an automated screening tool for gross motor development in early intervention, suitable for independently walking children aged one to six years old in Taiwan. The goal is to reduce the time cost of manual assessment and enable remote healthcare applications.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian willing to provide written informed consent.
* Males and females aged 1 to 6 years old.
* Capable of independent walking.

Exclusion Criteria:

- Non-native Chinese speakers.

Ages: 1 Year to 6 Years | Sex: All
Age Groups: Child
Study Population: Participants will be recruited from individuals referred for early intervention assessments at hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI-based gross motor development screening model compared to pediatric therapist's CDIIT gross motor subscale assessment | Day 1 (single assessment at enrollment).
  Accuracy will be calculated by comparing the AI model's classification results to pediatric therapists' assessments based on the CDIIT gross motor subscale.
  The accuracy formula is: (True Positive + True Negative) / Total number of cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes